CLINICAL TRIAL: NCT06960668
Title: Look at the Bright (Nature) Side: Improving Body Image and Associated Protective Factors and Reducing Body Image Threats With the Nature for Body Image (NBI) Project
Brief Title: Nature for Body Image
Acronym: NBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Silvia Cerea, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1216-a
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Body Image; Eating Behaviors; Self-Compassion; Interoception
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Nature Exposure (Experimental): The structured nature exposure sessions will be conducted twice a week, each lasting 30 minutes. Activities will include meditation, body scans, and grounding exercises in a natural setting (e.g., in a public park).
  Interventions: Behavioral: Nature for Body Image
- Simple Nature Exposure (Active Comparator): The simple nature exposure sessions will take place twice a week, with each session lasting 30 minutes. During these sessions, participants will spend time in nature (e.g., in a public park) without receiving specific instructions or guidance.
  Interventions: Behavioral: Simple nature exposure
- Structured Built Environment Exposure (Active Comparator): The structured built environment sessions will consist of five 30-minute sessions, mirroring the activities of the structured nature exposure sessions, but conducted entirely in non-natural settings.
  Interventions: Behavioral: Structured Built Environment Exposure

INTERVENTIONS:
Behavioral: Nature for Body Image — The intervention will include a range of activities in nature (e.g., in a public park), such as meditation, body scans, and grounding exercises.
  Arms: Structured Nature Exposure
Behavioral: Simple nature exposure — The intervention will simply involve spending time in nature (e.g., in a public park), without specific guidelines.
  Arms: Simple Nature Exposure
Behavioral: Structured Built Environment Exposure — The intervention will mirror the activities of the structured nature exposure intervention (e.g., meditation, body scans, and grounding exercises), but without any exposure to nature.
  Arms: Structured Built Environment Exposure

SUMMARY:
Nature exposure has been found to be particularly beneficial for body image, as recent studies have identified a positive association between time spent in nature and positive body image. Positive body image, defined as the ability to accept and respect one's body, has been linked to greater life satisfaction and engagement in healthy behaviors. Conversely, negative body image is recognized as a public health concern due to its detrimental effects on both physical and mental health. It has been associated with symptoms of Body Image Disorders (BIDs), including Eating Disorders (EDs) and Body Dysmorphic Disorder (BDD).

The Nature for Body Image (NBI) project aimed to examine the impact of a structured nature exposure intervention on improving body image among young women aged 18-35 years.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18-35 years old

Exclusion Criteria:

* Full-blown body image disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Negative Body Image | 5 weeks
  Assessed with the Italian - Body Image Concern Inventory (I-BICI), a 19-item self-report questionnaire measuring negative body image. Scores range from 19 to 95, with higher scores indicating greater negative body image.
Body Appreciation | 5 weeks
  Assessed with the Body Appreciation Scale-2 (BAS-2), a 10-item self-report questionnaire measuring body appreciation. Scores range from 10 to 50, with higher scores indicating greater body appreciation.
Functionality appreciation | 5 weeks
  Assessed with the Functionality Appreciation Scale (FAS), a 7-item self-report questionnaire measuring functionality appreciation. Scores range from 7 to 35, with higher scores indicating greater functionality appreciation.

SECONDARY OUTCOMES:
Dysfunctional Eating Behaviours and Risk of Developing Eating Disorders | 5 weeks
  Assessed with the Eating Disorder Risk Composite Score (EDRC) of the Eating Disorder Inventory-3 (EDI-3). The Eating Disorder Risk Composite Score (EDRC) investigates the risk of developing eating disorders with 25 items. Scores range from 0 to 100, with higher scores indicating greater risk of developing eating disorders.
Functional Eating Behaviors | 5 weeks
  Assessed with the Intuitive Eating Scale-2 (IES-2), a 23-item self-report questionnaire measuring intuitive eating. Scores range from 23 to 115, with higher scores indicating greater intuitive eating.
Embodiment | 5 weeks
  Assessed with the Experience of Embodiment Scale (EES), a 34-item self-report questionnaire measuring embodiment. Scores range from 34 to 170, with higher scores indicating greater embodiment.
Interoceptive Awareness | 5 weeks
  Assessed with the Multidimensional Assessment of Interoceptive Awareness (MAIA), a 32-item self-report questionnaire measuring interoceptive awareness. Scores range from 0 to 160, with higher scores indicating greater interoceptive awareness.
Self-compassion | 5 weeks
  Assessed with the Self-Compassion Scale (SCS), a 26-item self-report questionnaire measuring self-compassion. Scores range from 26 to 130, with higher scores indicating greater self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Psychology, University of Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No